CLINICAL TRIAL: NCT06252168
Title: Registry of Acute Myocardial Infarction
Acronym: RAMI-Tomsk
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: CRI-211
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction, Acute
Keywords: Acute Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Registry of Acute Myocardial Infarction (RAMI) aims at regular and centralized acquiring and processing standard information about verified and suspected cases of acute myocardial infarction (AMI), monitoring of AMI cases, and establishing AMI diagnosis based on standard diagnostic criteria by doctors involved in the registry. The RAMI obtains data from all medical institutions, which could potentially document any cases of suspected AMI.

DETAILED DESCRIPTION:
The study implements the methodology recommended by the World Health Organization (WHO) using unified diagnostic criteria (clinical, biochemical, electrocardiographic, and autopsy) for acute myocardial infarction (AMI). All primary information is recorded in a special primary registration card, which has been subject to updates in accordance with the requirements. All accumulated data is stored in RAMI analytic database. The database is designed and developed specifically for recording, accumulating, archiving, and statistical processing of collected data. It is equipped with a web user interface, a universal environment for generating consolidated distribution reporting, and the ability to import analytical data into expert analytical systems produced by other manufacturers. Data storage is implemented using the Oracle database management system. The information and analytical system of RAMI has passed the procedure of state registration of the database. Each reported case after the first 28 days from disease onset is assigned a specific diagnostic category (definite myocardial infarction, possible myocardial infarction, unconfirmed myocardial infarction, and insufficient data). At the end of each year of study, RAMI team calculates and analyzes the main epidemiological parameters, characterizing the disease distribution in the studied population (the city of Tomsk, Russian Federation) including morbidity, mortality, and lethality (general, in-hospital, and pre-hospital).

ELIGIBILITY:
Inclusion Criteria:

* age of at least 20 years;
* being a resident or visitor of the city of Tomsk at a time of AMI onset;
* the presence of definite AMI or possible AMI. Definite AMI is diagnosed in the presence of characteristic ECG changes, regardless of clinical course and changes in serum enzymes; or the presence of typical pain syndrome, "ambiguous" ECG changes, and definite increase in the activity of serum enzymes i.e. exceeding the upper limit of normal by 25% or more; or macroscopically detected focus of myocardial necrosis and (or) fresh thrombotic occlusion of the coronary artery. Possible AMI is registered in the presence of typical pain syndrome with ambiguous ECG changes and an ambiguous (up to 25%) increase in the levels of serum enzymes; or the presence of obstruction in the lumen of at least one coronary artery by at least 50% and (or) the presence of a post-infarction scar in the myocardium with a diameter of 0.5 cm or more, while simultaneously excluding a non-coronary cause of death. In case of atypical clinical picture, ambiguous or absent ECG changes, when the enzyme levels are not determined or their activity does not reach a pathological level, AMI case is considered unconfirmed. In the absence of data that could confirm or not confirm AMI, the case is interpreted as "insufficient data"

Exclusion Criteria:

* none.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population icnludes all subjects with verified and suspected acute myocardial infarction (AMI) in the city of Tomsk (Russian Federation) regardless of disease treatment, outcome, and healthcare institution esablishing diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 97500 (Estimated)
Dates: Start 1984-01-01 (Actual); Primary Completion 2049-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Early AMI lethality rate (%) | 28 days
  Early acute myocardial infarction (AMI) lethality rate is calculated as percentage (%) of fatal outcomes that occurred within 28 days since onset of disease among subjects with verified or suspected AMI.

SECONDARY OUTCOMES:
12-month AMI lethality rate (%) | 12 months
  12-month acute myocardial infarction (AMI) lethality rate is calculated as percentage (%) of fatal outcomes that occurred within one year since onset of disease among subjects with verified or suspected AMI.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei N. Repin, MD, PhD, Study Director — Tomsk NRMC; Sergey A. Okrugin, MD, PhD, Principal Investigator — Tomsk NRMC
Locations (1):
- Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No